CLINICAL TRIAL: NCT07179666
Title: Effectiveness of Neural Mobilization in Patients With Planter Fasciitis: A Pilot Study
Brief Title: Comparing Neural Mobilization and Traditional Physiotherapy in Plantar Fasciitis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-COHS-STD-137-Mar-2025
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Plantar Fasciitis
Keywords: neural moblization; conventional treatment
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural Mobilization Therapy (Experimental)
  Interventions: Other: Neural moblization group
- Conventional Physical therapy treatment (Experimental)
  Interventions: Other: Conventional therapy group

INTERVENTIONS:
Other: Neural moblization group — The intervention will involve neural mobilization of the tibial nerve, beginning with distal sliding through ankle dorsiflexion and foot eversion, followed by dorsiflexion of the toes. The movement will then be reversed into plantarflexion to allow proximal nerve excursion. In addition, a tensioner technique will be applied, in which participants will perform 45° hip flexion combined with ankle dorsiflexion and eversion, followed by knee extension, to place a controlled tensile load along the tibial nerve pathway.
  Arms: Neural Mobilization Therapy
Other: Conventional therapy group — The intervention will include manual therapy techniques such as myofascial release and soft tissue mobilization to reduce fascial tension and improve local circulation. Stretching exercises will be prescribed to target the plantar fascia, Achilles tendon, and gastrocnemius-soleus complex in order to enhance flexibility and reduce mechanical strain. In addition, ultrasound therapy will be utilized for its thermal and non-thermal effects to promote tissue healing and reduce inflammation.
  Arms: Conventional Physical therapy treatment

SUMMARY:
To evaluate the short-term effectiveness of neural mobilization targeting the posterior tibial nerve compared to traditional physiotherapy in cases diagnosed with plantar fasciitis, a pilot study will be conducted on 12 patients who will have been diagnosed with plantar fasciitis. Participants will be randomly divided into either the neural mobilization group or the conventional physiotherapy group, and all will receive three weeks of structured treatment. Results will be evaluated using techniques that will measure plantar pressure with Algometry, Foot Function Index (FFI) scores, and the Foot Health Status Questionnaire (FHSQ). Differences before and after treatment will be tested within the group using paired t-tests, and others will be examined between the groups with independent t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be selected within the age range of 19 to 40 years
* Meet the diagnostic criteria for plantar fasciitis, including symptoms of first-step pain in the morning and heel pain after long periods of standing, confirmed through clinical examination.

Exclusion Criteria:

* Individuals will be omitted from the study if they have undergone foot or ankle or foot surgery during the prior 12 months
* The presence of severe osteoarthritis, diabetic foot ulcers, or neuropathy

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-12 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Foot Function Index | 3 weeks
Foot Health Status Questionnaire | 3 weeks